CLINICAL TRIAL: NCT01410721
Title: Neural Markers and Rehabilitation of Executive Functioning in Veterans With TBI and PTSD
Brief Title: Neural Markers and Rehabilitation of Executive Functioning in Veterans With Traumatic Brain Injury and Posttraumatic Stress Disorder
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: United States Department of Defense (U.S. Federal Agency); Foundation of Hope, North Carolina (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 11-1292; PT100071 (Other: UNC)
Record Dates: First submitted 2011-08-03; First posted 2011-08-05 (Estimated); Last update posted 2018-12-13 (Actual); Status verified 2017-05

CONDITIONS: Traumatic Brain Injury; Posttraumatic Stress Disorder
Keywords: TBI; PTSD; Veterans
MeSH Terms: conditions — Brain Injuries, Traumatic; Stress Disorders, Post-Traumatic

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Cognitive Rehabilitation Intervention (Experimental): Baseline training and follow-up at two months and four months.
  Interventions: Behavioral: Cognitive Rehabilitation Intervention
- Cognitive Rehabilitation Control Arm (Active Comparator): Baseline training and follow-up at two months and four months.
  Interventions: Behavioral: Cognitive Rehabilitation Control Intervention

INTERVENTIONS:
Behavioral: Cognitive Rehabilitation Intervention — Baseline training and follow-up at two months and four months.
  Arms: Cognitive Rehabilitation Intervention
Behavioral: Cognitive Rehabilitation Control Intervention — Baseline training and follow-up at two months and four months.
  Arms: Cognitive Rehabilitation Control Arm

SUMMARY:
Up to half of all military service members with combat-related traumatic brain injury (TBI) also suffer from Posttraumatic Stress Disorder (PTSD). TBI and PTSD are each associated with cognitive problems in what are called 'executive functions' such as planning actions, inhibiting behavior, monitoring one's own thoughts and feelings, and solving problems day-to-day. These types of impairments occur more often among veterans with both TBI and PTSD than among those with only one of these conditions. The combination of TBI and PTSD in veterans has also been linked to problems with anger and violence, which are common complaints of veterans seeking mental health services post-deployment and have been shown to predict poor treatment outcomes in Iraq and Afghanistan veterans.

Although the relationship between combined TBI/PTSD diagnoses and post-deployment adjustment problems has been demonstrated, there has been little research into clinical interventions designed to reduce the severity of cognitive and affective symptoms in veterans with both TBI and PTSD. Therefore, the investigators propose a randomized clinical trial involving a cognitive rehabilitation intervention that targets improved executive functioning, with the participation of N=100 veterans diagnosed with both TBI and PTSD (n=50 in experimental group and n=50 comparison).

As part of the study, all participants will receive an iPod touch. Participants will be placed into one of the two study groups randomly. Based on which group participants are placed in, they will receive one of two different sets of iPod touch apps and programs that address and aim to improve different facets of cognitive functioning. Regardless of which group, Veterans will be instructed to daily practice iPod touch applications on cognitive functioning. Also, family members will be trained as "mentors" to reinforce use of the applications in everyday living environments. Trained facilitators will also travel to participants' homes to meet with veterans and family to observe behaviors in the home environment, arrive at strategies for applying new skills in their situations, troubleshoot any iPod technical problems, and review family mentoring processes.

The investigators will measure clinical outcomes using a comprehensive array of functional and structural methods at baseline and six months. The investigators hypothesize improved executive function among those in the experimental group as well as reduced irritability/impulsivity and improved social/occupational functioning. The investigators further hypothesize that, as a group, veterans participating in the cognitive rehabilitation program will show significant changes in neural activity associated with executive functions when comparing pre- and post-treatment EEG and fMRI responses.

Better understanding of the neural circuitry and neurocognitive function underlying executive function and associated affective control deficits in veterans with both TBI and PTSD, and how they relate to treatment outcome, will allow us to better identify therapeutic targets for cognitive rehabilitation. The current proposal aims to explore the relationship between brain function and connectivity in selective pathways/circuits, neuropsychological functioning, and cognitive rehabilitation response in veterans with both TBI and PTSD.

This study of the neurobiology and neuropsychology associated with intervention efficacy will allow us to identify veterans with both TBI and PTSD who are predisposed to positive treatment outcomes. To our knowledge, this will be the first attempt to integrate neurobiological and neurocognitive techniques with information about the efficacy of a theoretically and empirically driven cognitive rehabilitation intervention in veterans with combined TBI/PTSD diagnoses. This research may suggest additional avenues for assessment of clinical intervention efficacy and the identification of therapeutic targets (e.g. alteration of function in fronto-limbic circuits) relevant to the military population. Given links between TBI/PTSD, executive dysfunction, and anger, impulsivity, and aggression, efforts to rehabilitate cognitive function will be particularly important to ensure that current and future veterans adjust successfully when they return home to their families, workplaces, and communities.

DETAILED DESCRIPTION:
Background: It is estimated that up to half of all military service members with combat-related traumatic brain injury (TBI) also meet criteria for Posttraumatic Stress Disorder (PTSD). TBI and PTSD are both characterized by deficits in multiple cognitive domains, including attention, executive function, and affective and cognitive control. However, cognitive and affective sequelae associated with TBI are compounded by the presence of PTSD symptoms in returning veterans. Specifically, it has been shown that significant frontal lobe dysfunction, particularly disinhibition, occurs more often among veterans with both TBI and PTSD than among veterans diagnosed with only one of these conditions. The combination of TBI and PTSD in veterans has also been linked to problems with anger and violence, which are common complaints of veterans seeking mental health services post-deployment and have been shown to predict poor treatment outcomes in Iraq and Afghanistan veterans. Executive dysfunction, especially difficulty with attentional processing, is strongly related to hostility and aggressiveness in Iraq and Afghanistan veterans; increasingly so in the presence of TBI and PTSD.

Objective/Hypothesis: Although the relationship between combined TBI/PTSD diagnoses and post-deployment adjustment problems has been clearly demonstrated, there has been little empirical research into clinical interventions designed to reduce the severity of cognitive and affective symptoms in veterans with both TBI and PTSD. Therefore, the investigators propose to conduct a randomized trial of theoretically based cognitive rehabilitation to improve executive function and affective control among Iraq and Afghanistan veterans with both TBI and PTSD, and to measure clinical outcomes using a comprehensive array of functional and structural methods. The investigators hypothesize that improved executive function among those in the experimental group as well as reduced irritability/impulsivity and improved social/occupational functioning. The investigators further hypothesize that, as a group, veterans participating in the cognitive rehabilitation program will show significant changes in neural activity associated with executive functions when comparing pre- and post-treatment EEG and fMRI responses.

Specific Aims: Better understanding of the neural circuitry and neurocognitive function underlying executive function and associated affective control deficits in veterans with both TBI and PTSD, and how they relate to treatment outcome, will allow us to better identify therapeutic targets for cognitive rehabilitation. The current proposal aims to explore the relationship between brain function and connectivity in selective pathways/circuits, neuropsychological functioning, and cognitive rehabilitation response in veterans with both TBI and PTSD.

Study Design: Toward this end, the investigators propose a randomized clinical trial involving a cognitive rehabilitation intervention that targets improved executive functioning, with the participation of N=100 veterans diagnosed with both TBI and PTSD (n=50 in experimental group and n=50 receiving usual care). As part of the study, all participants will receive an iPod touch. Participants will be placed into one of the two study groups randomly. Based on which group participants are placed in, they will receive one of two different sets of iPod touch apps and programs that address and aim to improve different facets of cognitive functioning. Regardless of which group, Veterans will be instructed to daily practice iPod touch applications on cognitive functioning. Also, family members will be trained as "mentors" to reinforce use of the applications in everyday living environments. Trained facilitators will also travel to participants' homes to meet with veterans and family to review their respective applications and mentoring processes. The investigators will examine both cognitive and behavioral changes, as well as neural changes associated with cognitive rehabilitation using EEG and fMRI at baseline and six months.

Military Benefit: This study of the neurobiology and neuropsychology associated with intervention efficacy will allow us to identify veterans with both TBI and PTSD who are predisposed to positive treatment outcomes. To our knowledge, this will be the first attempt to integrate neurobiological and neurocognitive techniques with information about the efficacy of a theoretically and empirically driven cognitive rehabilitation intervention in veterans with combined TBI/PTSD diagnoses. This research may suggest additional avenues for assessment of clinical intervention efficacy and the identification of therapeutic targets (e.g. alteration of function in fronto-limbic circuits) relevant to the military population. Given links between TBI/PTSD, executive dysfunction, and anger, impulsivity, and aggression, efforts to rehabilitate cognitive function will be particularly important to ensure that current and future veterans adjust successfully when they return home to their families, workplaces, and communities.

ELIGIBILITY:
Inclusion Criteria:

OIF/OEF Veteran inclusion criteria include:

1. has served in one of the military branches (Army, Navy, Marines, Air Force, National Guard);
2. is between the ages of 18 and 65;
3. has served in Iraq or Afghanistan War since October 2001;
4. has screened positive for TBI and PTSD prior to baseline interview. Definition of TBI: The American Congress of Rehabilitation Medicine (ACRM) (Kay et al., 1993), Center for Disease Control (CDC, 2003), and Military TBI Task Force (http://www.div40.org/pdf/Military_TBI.pdf) have sought to define criteria for different types of head injuries. In the current DoD application, for both the research registry and pre-screening, criteria for TBI should be defined as a veteran who: 1. reports that during military service, head was hurt/injured in a way that caused problems; AND 2. endorses at least one of the following:

   * loss of consciousness or getting "knocked out."
   * immediately after the injury or upon regaining consciousness, being dazed or "seeing stars."
   * immediately after the injury or upon regaining consciousness, being unable to recall the event.
   * being over one hour after the injury was it before veteran started remembering new things again.
   * needing brain surgery after the injury.

Definition of PTSD: For the purposes of the current research, we use the Diagnostic Statistical Manual-IV-TD (DSM-IV-TR) definition of PTSD for the purposes of the current research. Specifically, subjects must report a traumatic event according to DSM criteria and report experiencing re-experiencing, avoidance, and hyperarousal symptoms to qualify for the diagnosis. Study registries define PTSD as having a score above the cut-off of 60 on the Clinical Assessment of PTSD (CAPS). We will re-screen potential participants before enrollment by administering the PTSD Checklist, scores above 50 indicative of PTSD among OIF/OEF veterans. Please note below that the CAPS will be administered as part of the main clinical interview after veterans have signed informed consent.

Family member inclusion criteria include: (1) has family member/friend who served in one of the military branches (Army, Navy, Marines, Air Force, National Guard); (2) age 18-65; and (3) has family member who served at least one tour in Iraq or Afghanistan since October 2001 and meets above criteria Inclusion of Women and Minorities in Study: It is anticipated that the distribution of our sample by gender and race/ethnicity will reflect the client population served by the North Carolina healthcare system. No one will be excluded from the study because of gender or racial/ethnic group.

Exclusion Criteria:

Since MRI sessions are a part of the study, subjects should not participant if:

1. They have any foreign metal objects or implants in their body as determined by the safety questionnaires.
2. Veteran is a woman and is pregnant or unwilling to take a pregnancy test.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 241 (Actual)
Dates: Start 2012-01; Primary Completion 2016-02 (Actual); Study Completion 2016-02 (Actual)

PRIMARY OUTCOMES:
Executive Function | 6 month
  Executive function is hypothesized to be improved in the experimental group, as evidenced by increased scores on neuropsychological measures from Dellis-Kaplan Executive Functioning System.

SECONDARY OUTCOMES:
Impulsivity | 6 months
  It is hypothesized that participants in the experimental group will shown reduced impulsivity, as measured by the Barrat Impulsivity Scale.
Interpersonal Conflict | 6 months
  It is hypothesized that participants in the experimental group will shown reduced interpersonal conflict, as measured by the Conflict Tactics Scale.

CONTACTS AND LOCATIONS:
Overall Officials: Eric B. Elbogen, Ph.D, Principal Investigator — UNC
Locations (1):
- UNC, Chapel Hill, North Carolina, United States

REFERENCES:
- [Derived] Elbogen EB, Dennis PA, Van Voorhees EE, Blakey SM, Johnson JL, Johnson SC, Wagner HR, Hamer RM, Beckham JC, Manly T, Belger A. Cognitive Rehabilitation With Mobile Technology and Social Support for Veterans With TBI and PTSD: A Randomized Clinical Trial. J Head Trauma Rehabil. 2019 Jan/Feb;34(1):1-10. doi: 10.1097/HTR.0000000000000435. PMID 30169439
- See also: Related publication — https://www.ncbi.nlm.nih.gov/pubmed/30169439